CLINICAL TRIAL: NCT04525560
Title: Efficacy, Safety and Tolerability of Different Bowel Preparation Before Colonoscopy in Children Over 2 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BP/2+
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Child Obesity; Bowel Preparation
Keywords: Child; Electronic colonoscopy; bowel preparation; polyethylene glycol with electrolyte solution
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-ELS-S (Experimental): The dosage of PEG-ELS is given according to body weight: 10-15 kg, PEG-ELS 0.75 L; 15-22.5 kg, PEG-ELS 1.5 L; 22.5-30 kg, PEG-ELS 2.25 L; more than 30 kg, PEG-ELS 3 L.
  Interventions: Other: PEG-ELS-S
- PEG-ELS-L (Active Comparator): The dosage of PEG-ELS is given according to body weight: 10-15 kg, PEG-ELS 0.75 L; 15-22.5 kg, PEG-ELS 1.5 L; 22.5-30 kg, PEG-ELS 2.25 L; more than 30 kg, PEG-ELS 3 L.
  Interventions: Other: PEG-ELS-L

INTERVENTIONS:
Other: PEG-ELS-S — 2/3 dose of PEG-ELS was taken orally from the evening on the day before colonoscopy, and the remaining 1/3 dose of PEG-ELS was orally administered in the morning of the next day.
  Arms: PEG-ELS-S
Other: PEG-ELS-L — PEG-ELS is given orally on the day before colonoscopy, which is divided into 10-12 portions and taken one portion every hour. If half of the total amount is not completed at afternoon ward round the day before colonoscopy, nasogastric feeding is recommended.
  Arms: PEG-ELS-L

SUMMARY:
Electronic colonoscopy plays an important role in the diagnosis and follow-up of intestinal diseases in children.

DETAILED DESCRIPTION:
The adequacy of bowel preparation before colonoscopy is particularly important for the visualization of intestinal mucosa under colonoscopy. Some studies have shown that bowel preparation must be customized according to the age, weight and clinical status of the child. However, there is no internationally recognized standard scheme for pediatric intestinal reserve. In pediatric clinical trials, polyethylene glycol with electrolyte solution (PEG-ELS) is more effective than bisacodyl, folium sennae and magnesium citrate. PEG-ELS is an electrolyte balanced isotonic solution, which can be used to clean the intestinal tract by large volume irrigation. Polyethylene glycol 4000 is a long-chain linear polymer, which can hardly absorb and decompose after oral administration. It can effectively increase the composition of intestinal fluid, stimulate intestinal peristalsis, cause watery diarrhea, and achieve the purpose of cleaning the intestine. The inorganic salt composition and proper amount of water in the formula ensure the balance of water and electrolyte exchange between intestinal tract and body fluid. In this study, PEG-ELS short protocol and long protocol were selected for intestinal preparation, and the effectiveness and safety of different intestinal preparation protocols under electronic colonoscopy for children over 2 years old were compared.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed children in Department of Gastroenterology at Children's Hospital of Fudan University
* According to the indications of electronic colonoscopy, colonoscopy was performed for the first time
* Age: 2-22 years old

Exclusion Criteria:

* Having contraindications of electronic colonoscopy
* Having contraindications of general anesthesia
* Previous abdominal surgery
* Chronic constipation
* There is evidence of intestinal stenosis and gastrointestinal malformation
* Laxatives or drugs in the intestinal preparation protocol of this study have been used before bowel preparation
* Disagree the use of the bowel preparation protocol developed in the study

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 315 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing | During the operation of electronic colonoscopy (about 15 min )
  Bowel cleansing was assessed by Boston bowel preparation scale (BBPS). The scores of left, middle and right colon were added up to the total score of BBPS, with the lowest score of 0 and the highest score of 9. The score of 8-9 represents excellent bowel preparation, 6-7 represents good, 4-5 represents average, and 0-3 represents poor. Excellent and good for intestinal preparation are qualified, general and poor for intestinal preparation are unqualified.

SECONDARY OUTCOMES:
Compliance with polyethylene glycol with electrolyte solution (PEG-ELS) | During bowel preparation (about 24 hours)
  This variable is a binary variables (good/poor). Poor compliance was defined as PEG-ELS dosage less than 75% of the prescribed dose. Good compliance was defined as PEG-ELS dosage more than 75% of the prescribed dose. Prescribed dose and actually oral dose were recorded by nurse.
Adverse reactions receiving polyethylene glycol with electrolyte solution | During bowel preparation (about 24 hours)
  This variable is a binary variables (Yes/No). The variable would be set to "Yes" as any adverse reactions including Nausea, vomiting, abdominal distension, abdominal pain or allergic to PEG-ELS appeared during bowel preparation.
Rate of nasal feeding PEG-ELS | During bowel preparation (about 24 hours)
  Rate of nasal feeding PEG-ELS. Nasogastric feeding is recommended for those who cannot complete the prescribed amount.
Enema rate before colonoscopy | immediately before colonoscopy
  At 8 am on the day of electronic colonoscopy, no food and water were given from 8 am. At 11 am on the day of colonoscopy, the last assessment of stool was conducted. If the Bristol stool form scale (BSFS) ≤ 5 points, colonoscopy should be cancelled and bowel preparation time should be prolonged; if BFSF = 6 points, Warm normal saline (50 ml/kg) was given for enema; if BFSF = 7 points, no enema.
Times of washing under colonoscopy | During the operation of electronic colonoscopy (about 15 mins)
  If the visual field is not clear, it should be washed during the operation of electronic colonoscopy.
Adverse events | up to 30 minutes after colonoscopy
  It is a repeated measured variable. This variable is a binary variables (Yes/No). The variable would be set to "Yes" as any adverse reactions. An adverse event refers to the event that occurs after a patient in a clinical study accepts a research-based product, which does not necessarily have a causal relationship with the test product. Adverse events are diseases, signs or symptoms (including abnormal laboratory results) that occur or worsen during the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No